CLINICAL TRIAL: NCT06327503
Title: Salivary Signal Molecules Relevant for Neural and Vascular Homeostasis in Patients With Type 2 Diabetes Mellitus
Brief Title: Salivary Signal Molecules for Neural and Vascular Homeostasis in T2DM
Status: Completed | Type: Observational
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Marija S. Milic, Assistant Professor, University of Belgrade
Other Study IDs: 36/7-2024
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of unstimulated whole saliva kept on -80 Celsius degrees until laboratory analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T2DM patients: patients with diagnosed controlled Type 2 Diabetes Mellitus with or without systemic complications
  Interventions: Other: saliva samples collecting
- non-T2DM patients: age and general health matched control group without Type 2 Diabetes Mellitus
  Interventions: Other: saliva samples collecting

INTERVENTIONS:
Other: saliva samples collecting — non-invasive collection of unstimulated whole saliva by spitting method into sterile plastic container

SUMMARY:
Various signal molecules are detected in blood and tissues of patients with T2DM, that are important for the function of neural tissue in diabetic setting. Among them, specifically important are neuroprotective and neurotrophic growth factors such as nerve growth factor (NGF), glial cells - derived neurotrophic factor (GDNF) and brain-derived neurotrophic factor (BDNF). Furthermore, several other signal molecules are discovered to affect vascular tissues homeostasis in T2DM, including soluble alpha-klotho (s-Klotho), vascular endothelial growth factor (VEGF) and interleukin-6 (IL-6). Most of these molecules are also detected in saliva in various states and diseases of orofacial system, but data about their levels in saliva of T2DM patients are lacking, although neural and vascular diabetic complications are present in orofacial tissues and organs. Also, there is no data about presence and levels of s-Klotho in saliva of healthy or T2DM patients, although it was reported that this molecule exerts protective effect on the salivary glands tissue. Salivary opiorphin is recently discovered pentapeptide, primarily isolated from saliva. It acts as an inhibitor of the enzymes that perform degradation of endogenous antinociceptive molecules enkephalins, affecting nociceptive signal transduction. This may be of special importance since some intraoral complications of T2DM (e.g. burning mouth) may have underlying peripheral neural changes as a pathophysiological mechanism. Against this background, the aim of the study is to detect the presence and levels of mentioned signal molecules in saliva of patients with and without T2DM.

ELIGIBILITY:
Inclusion Criteria:

* patients with maxillary and mandibular total edentulism with and without T2DM
* for patients with T2DM - presence of controlled T2DM

Exclusion Criteria:

* presence of the acute pain or swelling in orofacial region
* antibiotic therapy up to three weeks prior to study start
* conditions or diseases that affect the function of salivary glands (e.g. Sjogren syndrome)
* radiotherapy of the orofacial region
* tobacco smokers
* alcohol and/or drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will comprise age and general health matched groups with and without T2DM, with total edentulism in the upper and lower jaw
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
NGF levels in saliva | on 5th day after sample collection
  levels of nerve growth factor in saliva samples obtained from T2DM and non-T2DM groups, detected by means of ELISA method
GDNF levels in saliva | on 5th day after sample collection
  levels of glial-cells derived neurotrophic factor in saliva samples obtained from T2DM and non-T2DM groups, detected by means of ELISA method
BDNF levels in saliva | on 5th day after sample collection
  levels of brain derived neurotrophic factor in saliva samples obtained from T2DM and non-T2DM groups,
s-Klotho levels in saliva | on 5th day after sample collection
  levels of soluble alpha-klotho in saliva samples obtained from T2DM and non-T2DM groups,
VEGF levels in saliva | on 5th day after sample collection
  levels of vascular endothelial growth factor in saliva samples obtained from T2DM and non-T2DM groups,
IL-6 levels in saliva | on 5th day after sample collection
  levels of interleukin-6 in saliva samples obtained from T2DM and non-T2DM groups,
opiorphin levels in saliva | on 5th day after sample collection
  levels of opiorphin in saliva samples obtained from T2DM and non-T2DM groups,

SECONDARY OUTCOMES:
unstimulated saliva flow | immediately after sample collection
  measuring of the flow of unstimulated saliva by dividing the volume of saliva with the time necessary for the sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Marija S Milic, DDS PhD, Principal Investigator — University of Belgrade School of Dental Medicine
Locations (1):
- University of Belgrade School of Dental Medicine, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP